CLINICAL TRIAL: NCT00025727
Title: A Phase III, Randomized, Multicenter, Parallel Group, Open-Label, Three Arm Study to Compare the Efficacy and Safety of Two Dosing Regimens of GW433908/Ritonavir (700mg/100mg Twice Daily or 1400mg/200mg Once Daily) Versus Lopinavir/Ritonavir (400mg/100mg Twice Daily) for 48 Weeks in Protease Inhibitor Experienced HIV-Infected Adults Experiencing Virological Failure
Brief Title: Comparison of Two Dosing Regimens of GW433908/Ritonavir Versus Lopinavir/Ritonavir for 48 Weeks in HIV Patients Who Have Taken Protease Inhibitors and Experienced Virological Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GlaxoSmithKline (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 316C
Record Dates: First submitted 2001-10-15; First posted 2001-10-16 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-06

CONDITIONS: HIV Infections
Keywords: HIV-1; HIV Protease Inhibitors; Ritonavir; RNA, Viral; Anti-HIV Agents; Viral Load; ABT 378; VX-175
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir; fosamprenavir

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Ritonavir
Drug: GW433908

SUMMARY:
The purpose of this study is to test 2 different dosing regimens of GW433908/ritonavir (RTV) versus lopinavir (LPV)/RTV when each is given with 2 active reverse transcriptase inhibitors (RTIs), in patients who have taken anti-HIV drugs without success.

DETAILED DESCRIPTION:
Patients will receive 2 dosing regimens of GW433908/RTV or LPV/RTV, in combination with 2 active RTIs, after failing their first or second protease inhibitor-containing regimen. Patients are required to be on therapy at time of screening and must remain on this therapy until Day 1.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have a viral load of 1,000 or more copies/ml.
* Have taken protease inhibitors (PIs).
* Have taken PI drugs for at least 12 straight weeks and have had virologic failure on the PIs.
* Are now taking antiretroviral therapy.
* Are male or female and are at least 13 years old (or 18 if local requirement) and can provide consent from parent or guardian if under 18.
* Are females unable to have children or, if are able to have children, are not pregnant and agree to use approved birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken APV or LPV for more than 1 week.
* Have taken tenofovir disoproxil fumarate (TDF) or adefovir.
* Have taken more than 2 PIs.
* Are unable to take 2 active RTIs, as specified by the study.
* Have an active CDC Category C disease.
* Have certain abnormal laboratory tests.
* Are pregnant or breast-feeding.
* Have a serious health problem (e.g., diabetes, heart problems, hepatitis) that might risk the safety of the patient.
* Have a history of significant kidney or bone disease.
* Are not able to take drugs by mouth and cannot absorb them.
* Have had pancreatitis or hepatitis within the previous 6 months.
* Have a drug allergy or other allergy which might cause a problem during the study.
* Have had radiation or chemotherapy within 28 days of taking the study drug, or expect to need these during the study.
* Have taken drugs that affect the immune system (corticosteroids, interleukins, interferons) or drugs with anti-HIV activity (hydroxyurea or foscarnet) within 28 days prior to taking the study drug.
* Have had any HIV vaccine within 3 months before taking the study drug.
* Have taken certain other drugs within 28 days prior to taking the study drug, or expect to need them during the study.
* Use alcohol or illicit drugs in a way that the doctor feels would interfere with the study.
* Are not able to take the study drugs.
* Have inadequate kidney function.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330
Dates: Start 2001-05

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Phoenix Body Positive, Phoenix, Arizona
  - Ocean View Internal Medicine, Long Beach, California
  - Bisher Akil, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - Orange Coast Med Group, Newport Beach, California
  - Pacific Horizons Med Group, San Francisco, California
  - Denver Inf Disease Consultants, Denver, Colorado
  - Physicans Home Service, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Bach and Godofsky, Bradenton, Florida
  - Community Health Care, Fort Lauderdale, Florida
  - Therafirst Med Ctr, Fort Lauderdale, Florida
  - North Broward Hosp District / HIV Clinical Research, Fort Lauderdale, Florida
  - Florida ID Group, Orlando, Florida
  - Discovery Alliance Inc, Pensacola, Florida
  - West Florida Clinical Research Ctr, Pensacola, Florida
  - Med College of Georgia, Augusta, Georgia
  - Rush Med College / Dept of Infectious Diseases, Chicago, Illinois
  - Boston Med Ctr / Evans - 556, Boston, Massachusetts
  - Abbott-Northwestern Hosp / Clinic 42, Minneapolis, Minnesota
  - Southampton Healthcare Inc, St Louis, Missouri
  - South Jersey Infectious Diseases Inc, Somers Point, New Jersey
  - ID Care Inc, Somerville, New Jersey
  - Garden State Infectious Diseases / E I P Kennedy Health Sys, Voorhees Township, New Jersey
  - Gervais Frechette, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Summa Health System, Akron, Ohio
  - Fanno Creek Clinic, Portland, Oregon
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Methodist Healthcare, Memphis, Tennessee
  - Joseph Gathe, Houston, Texas
  - Virginia Commonwealth Univ, Richmond, Virginia